CLINICAL TRIAL: NCT00852761
Title: A Study to Evaluate Safety and Efficacy of Clobetasol Propionate for Treatment of Plaque-Type Psoriasis in Adult Subjects.
Brief Title: A Study to Evaluate the Efficacy and Tolerability of Topical Therapies for the Condition of Plaque-Type Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114569; U0280-402
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Plaque-Type Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Clobetasol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olux-E Foam (Experimental): Olux-E (clobetasol propionate 0.05%) foam
  Interventions: Drug: Olux-E Foam
- Clobex lotion (Active Comparator): Clobex (clobetasol propionate 0.05%) lotion.
  Interventions: Drug: Clobex lotion

INTERVENTIONS:
Drug: Olux-E Foam — Olux-E (clobetasol propionate 0.05%) foam. Starting at baseline, subjects were to apply twice daily Olux-E foam to the affected elbows and/or knees up to day 15.
  Arms: Olux-E Foam
Drug: Clobex lotion — Clobetasol propionate 0.05% lotion. Starting at baseline, subjects were to apply twice daily Clobex lotion to the affected elbows and/or knees up to day 15
  Other Names: clobetasol lotion; Clobex
  Arms: Clobex lotion

SUMMARY:
The purpose of the study is to determine the efficacy and safety of two different forms of a topical steroid (clobetasol propionate) in patients with plaque-type psoriasis.

DETAILED DESCRIPTION:
This study is being conducted to obtain efficacy and tolerability data for two clobetasol propionate therapies in the treatment of plaque-type psoriasis. Subjects will be randomized to only one of the two therapies for treatment throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body surface area (BSA) affected with psoriasis between 4% and 20% .
* Target lesion of at least 2 cm² on the elbow and/or knee, with a score of 2 or 3 on the Psoriasis Grading Scale for Target Lesion.
* Elbow and/or knee plaque-type psoriasis with a Psoriasis Global Assessment of mild or moderate (2 or 3).
* Definitive diagnosis of elbow and/or knee plaque-type psoriasis.
* Capable of understanding and willing to provide a signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol-specific procedures were performed.
* Male or female, 18 years of age or older at the time that the consent form was signed.
* Able to complete the study and comply with study instructions.
* Female subjects of childbearing potential must have had a negative pregnancy test. Sexually active women of childbearing potential participating in the study must have been using a medically acceptable form of contraception.

Exclusion Criteria:

* Use of any emollient applied to psoriasis plaques treated with the study medication during the study.
* Other serious skin disorder or any chronic medical condition that is not well controlled.
* Female subjects who are pregnant, trying to become pregnant or lactating.
* Any major illness within 30 days prior to the baseline visit.
* Received any investigational drug or treatment within 30 days of the baseline visit or who are scheduled to receive an investigational drug or treatment other than the study products during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical research center
Groups:
- Olux-E Foam: Olux-E (Clobetasol propionate 0.05 percent) foam. Administered twice daily to the elbow and/or knees, morning and evening, after washing with a mild cleanser.
- Clobex Lotion: Clobex (Clobetasol propionate 0.05 percent) lotion. Administered twice daily to the elbow and/or knees, morning and evening, after washing with a mild cleanser.
Period: Overall Study
Arm/Group | Olux-E Foam | Clobex Lotion
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olux-E Foam | Clobex Lotion | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Customized [Mean (Standard Deviation); unit: years] | 48.2 (11.7) | 48.6 (13) | 48.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women and is measured in kg/m^2.
  kg/m^2 | 31.2 (6.4) | 30.0 (8.8) | 30.6 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: At Least a One Grade Improvement for the Target Psoriasis Lesion on the Elbow or Knee (Psoriasis Grading Scale)
Description: Number of participants who achieved a minimum 1-grade improvement in elbow and/or knee lesion using the Psoriasis Grading Scale for Target Lesion Score: 0 = No evidence of scaling, erythema, or elevation. 1 = Minimal; occasional scale, faint erythema, slight elevation. 2 = Mild; fine scales, light red color, slight elevation. 3 = Moderate; coarse scales, moderate red coloration and elevation . 4 = Marked; thick scale, bright red coloration, marked elevation. 5 = Severe; very thick tenacious scale predominates, dusky to deep red coloration, very marked elevation.
Time Frame: Baseline to day 15
Population: ITT
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants | 15 | 14

2. Secondary Outcome: At Least 1 Grade Improvement Psoriasis Grading Scale
Description: Number of participants who achieve a minimum one grade improvement or more in their elbow and/or knee target lesion as defined by the Psoriasis Grading Scale for Target Lesion.
  The scale is the same as used for the primary outcome (0 through 5).
Time Frame: Baseline, days 3 and 8
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 3 | 9 | 10
  Day 8 | 14 | 14
Statistical Analysis 1: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.7298, Chi-squared — This is the result for the Day 3 analysis
Statistical Analysis 2: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 1.0000, Chi-squared — This is the result for the Day 8 analysis

3. Secondary Outcome: At Least a 2 Grade Improvement Psoriasis Grading Scale
Description: Number of participants who achieve a minimum two grade improvement or more in their elbow and/or knee target lesion as defined by the Psoriasis Grading Scale for Target Lesion.
  The scale is the same as used for the primary outcome (0 through 5).
Time Frame: Baseline, days 3, 8, 15
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 3 | 2 | 1
  Day 8 | 5 | 13
  Day 15 | 5 | 13
Statistical Analysis 1: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.7298, Chi-squared — This is the result for the Day 3 analysis
Statistical Analysis 2: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.0060, Chi-squared — This is the result for the Day 8 analysis
Statistical Analysis 3: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.0060, Chi-squared — This is the result for the Day 15 analysis

4. Secondary Outcome: At Least a 3 Grade Improvement Psoriasis Grading Scale
Description: Number of participants who achieve a minimum of three grade improvement or more in their elbow and/or knee target lesion as defined by the Psoriasis Grading Scale for Target Lesion.
  The scale is the same as used for the primary outcome (0 through 5).
Time Frame: Baseline, days 3, 8, 15
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 8 | 0 | 2
  Day 15 | 0 | 4
Statistical Analysis 1: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.0332, Chi-squared — Data apply to Day 15

5. Secondary Outcome: At Least 1 Grade Improvement in the Psoriasis Global Assessment
Description: Number of participants who acheive at least a 1 grade improvement in the Psoriasis Global Assessment. 0 = Clear; 1 = Almost Clear; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Baseline, days 3, 8, 15
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 3 | 6 | 7
  Day 8 | 10 | 13
  Day 15 | 14 | 14

6. Secondary Outcome: At Least a 2 Grade Improvement in the Psoriasis Global Assessment
Description: Number of participants who acheive at least a 2 grade improvement in the Psoriasis Global Assessment. 0 = Clear; 1 = Almost Clear; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Baseline, days 3, 8, 15
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 3 | 0 | 1
  Day 8 | 6 | 7
  Day 15 | 3 | 10
Statistical Analysis 1: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.3101, Chi-squared — This is the result for the Day 3 analysis
Statistical Analysis 2: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.7242, Chi-squared — This is the result for the Day 8 analysis
Statistical Analysis 3: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.0135, Chi-squared — This is the p value for day 15

7. Secondary Outcome: At Least a 3 Grade Improvement in the Psoriasis Global Assessment
Description: Number of participants who acheive at least a 3 grade improvement in the Psoriasis Global Assessment. 0 = Clear; 1 = Almost Clear; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Baseline, days 3, 8, 15
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 3 | 0 | 0
  Day 8 | 0 | 0
  Day 15 | 0 | 3

8. Secondary Outcome: At Least 1 Grade Improvement in Subject's Global Assessment
Description: Number of participants who achieve treatment success (minimum one grade improvement or more) in their elbow and/or knee target lesion as defined by the Subject's Global Assessment. 0 = My skin is completely clear, except for residual hyperpigmentation. 1 = My psoriasis is almost clear; patchy fine scaling may be present. 2 = My psoriasis is mild, with a small amount of psoriasis. 3 = My psoriasis is moderate, between slight and definitely noticeable. 4 = My psoriasis is very noticeable. 5 = My psoriasis is severe with severe redness, thick scaling, plaques.
Time Frame: Baseline, days 3, 8, 15
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 3 | 8 | 12
  Day 8 | 15 | 16
  Day 15 | 15 | 17
Statistical Analysis 1: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.1449, Chi-squared — P value at day 15
Statistical Analysis 2: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.1634, Chi-squared — P value at day 3
Statistical Analysis 3: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.5454, Chi-squared — P value at day 8

9. Secondary Outcome: At Least a 2 Grade Improvement in Subject's Global Assessment
Description: Number of participants who achieve treatment success (minimum two grade improvement or more) in their elbow and/or knee target lesion as defined by the Subject's Global Assessment. 0 = My skin is completely clear, except for residual hyperpigmentation. 1 = My psoriasis is almost clear; patchy fine scaling may be present. 2 = My psoriasis is mild, with a small amount of psoriasis. 3 = My psoriasis is moderate, between slight and definitely noticeable. 4 = My psoriasis is very noticeable. 5 = My psoriasis is severe with severe redness, thick scaling, plaques.
Time Frame: Baseline, days 3, 8, 15
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 3 | 4 | 3
  Day 8 | 10 | 11
  Day 15 | 13 | 14
Statistical Analysis 1: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.6715, Chi-squared — This is the p value for day 15
Statistical Analysis 2: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.7242, Chi-squared — This is the p value for day 8
Statistical Analysis 3: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.6715, Chi-squared — This is the p value for day 3

10. Secondary Outcome: At Least a 3 Grade Improvement in Subject's Global Assessment
Description: Number of participants who achieve treatment success (minimum three grade improvement or more) in their elbow and/or knee target lesion as defined by the Subject's Global Assessment. 0 = My skin is completely clear, except for residual hyperpigmentation. 1 = My psoriasis is almost clear; patchy fine scaling may be present. 2 = My psoriasis is mild, with a small amount of psoriasis. 3 = My psoriasis is moderate, between slight and definitely noticeable. 4 = My psoriasis is very noticeable. 5 = My psoriasis is severe with severe redness, thick scaling, plaques.
Time Frame: Baseline, days 3, 8, 15
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 3 | 0 | 0
  Day 8 | 6 | 8
  Day 15 | 8 | 11
Statistical Analysis 1: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.4858, Chi-squared — P value on day 8
Statistical Analysis 2: Comparison: Olux-E Foam vs Clobex Lotion; Test type: Superiority or Other; p = 0.3001, Chi-squared — P value on day 15

11. Secondary Outcome: Median Change in Psoriasis Grading Scale
Description: Median improvement in elbow and/or knee lesion using the Psoriasis Grading Scale for Target Lesion Score: 0 = No evidence of scaling, erythema, or elevation. 1 = Minimal; occasional scale, faint erythema, slight elevation. 2 = Mild; fine scales, light red color, slight elevation. 3 = Moderate; coarse scales, moderate red coloration and elevation . 4 = Marked; thick scale, bright red coloration, marked elevation. 5 = Severe; very thick tenacious scale predominates, dusky to deep red coloration, very marked elevation.
Time Frame: Baseline, Days 3, 8, 15
Population: ITT
Measure: Median (Inter-Quartile Range); unit: unites on a scale
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
unites on a scale
  Day 3 | -1 [-1 to 0] | -1 [-1 to 0]
  Day 8 | -1 [-2 to -1] | -2 [-2 to -1]
  Day 15 | -1 [-2 to -1] | -2 [-2 to -2]

12. Secondary Outcome: Dermatology Quality of Life - Symptoms and Feelings
Description: Dermatology Quality of Life (DLQI) measures quality of life for people with skin conditions.
  Sum of scores for questions 1 and 2. Score range from 0 to 6. A higher score denotes a more impaired quality of life
Time Frame: Baseline, Days 3, 8, 15
Population: ITT (Note: some subjects did not complete the survey at all timepoints; however, all data available was analyzed.)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
units on a scale
  Day 3, n=16, 17 | 1.94 (1.12) | 2.41 (1.70)
  Day 8, n=17, 17 | 1.06 (1.2) | 1.35 (1.32)
  Day 15, n=17, 17 | 0.82 (0.95) | 0.94 (1.14)

13. Secondary Outcome: Dermatology Quality of Life - Daily Activities
Description: Dermatology Quality of Life (DLQI) measures quality of life for people with skin conditions.
  Sum of scores for questions 3 and 4. Score range from 0 to 6. A higher score denotes a more impaired quality of life
Time Frame: Baseline, Days 3, 8, 15
Population: ITT (Note: some subjects did not complete the survey at all timepoints; however, all data available was analyzed.)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
units on a scale
  Day 3, n=16, 17 | 0.56 (0.96) | 1.41 (1.23)
  Day 8, n=17, 17 | 0.53 (0.94) | 0.88 (1.05)
  Day 15, n=17, 17 | 0.53 (1.07) | 0.82 (1.29)

14. Secondary Outcome: Dermatology Quality of Life - Leisure
Description: Dermatology Quality of Life (DLQI) measures quality of life for people with skin conditions.
  Sum of scores for questions 5 and 6. Score range from 0 to 6. A higher score denotes a more impaired quality of life
Time Frame: Baseline, Days 3, 8, 15
Population: ITT (Note: some subjects did not complete the survey at all timepoints; however, all data available was analyzed.)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
units on a scale
  Day 3, n=16, 17 | 0.5 (0.97) | 0.94 (1.30)
  Day 8, n=17, 17 | 0.47 (0.94) | 0.41 (0.87)
  Day 15, n=17, 17 | 0.35 (1.0) | 0.24 (0.56)

15. Secondary Outcome: Dermatology Quality of Life - Work and School
Description: Dermatology Quality of Life (DLQI) measures quality of life for people with skin conditions.
  Sum of scores for questions 7. Score range from 0 to 3. A higher score denotes a more impaired quality of life
Time Frame: Baseline, Days 3, 8, 15
Population: ITT (Note: some subjects did not complete the survey at all timepoints; however, all data available was analyzed.)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
units on a scale
  Day 3, n=15, 17 | 0.13 (0.35) | 0.24 (0.56)
  Day 8, n=16, 17 | 0.06 (0.25) | 0.12 (0.33)
  Day 15, n=17, 17 | 0.06 (0.24) | 0.06 (0.24)

16. Secondary Outcome: Dermatology Quality of Life - Personal Relationships
Description: Dermatology Quality of Life (DLQI) measures quality of life for people with skin conditions.
  Sum of scores for questions 8 and 9. Score range from 0 to 6. A higher score denotes a more impaired quality of life
Time Frame: Baseline, Days 3, 8, 15
Population: ITT (Note: some subjects did not complete the survey at all timepoints; however, all data available was analyzed.)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
units on a scale
  Day 3, n=15, 17 | 0.33 (0.49) | 0.41 (0.80)
  Day 8, n=16, 17 | 0.25 (0.45) | 0.29 (0.77)
  Day 15, n=17, 17 | 0.18 (0.53) | 0.12 (0.33)

17. Secondary Outcome: Dermatology Quality of Life - Treatment
Description: Dermatology Quality of Life (DLQI) measures quality of life for people with skin conditions.
  Sum of scores for question 10. Score range from 0 to 3. A higher score denotes a more impaired quality of life
Time Frame: Baseline, Days 3, 8, 15
Population: ITT (Note: some subjects did not complete the survey at all timepoints; however, all data available was analyzed.)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
units on a scale
  Day 3, n=16, 17 | 0.31 (0.60) | 0.35 (0.61)
  Day 8, n=17, 17 | 0.29 (0.59) | 0.24 (0.44)
  Day 15, n=17, 17 | 0.18 (0.39) | 0.24 (0.44)

18. Secondary Outcome: Total Dermatology Life Quality Index (DLQI) Score
Description: Dermatology Quality of Life (DLQI) measures quality of life for people with skin conditions.
  Sum of scores for all questions. Score range from 0 to 30. A higher score denotes a more impaired quality of life
Time Frame: Baseline, Days 3, 8, 15
Population: ITT (Note: some subjects did not complete the survey at all timepoints; however, all data available was analyzed.)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
units on a scale
  Day 3 | 3.75 (2.82) | 5.76 (4.64)
  Day 8 | 2.65 (3.44) | 3.29 (3.64)
  Day 15 | 2.12 (3.64) | 2.41 (3.00)

19. Secondary Outcome: Dermatology Life Quality Index (DLQI) Categories
Description: Number of participants who indicated one of the following for total DLQI: 0-1 No effect on the patient's life; 2-5 Small effect on the patient's life; 6-10 Moderate effect on the patient's life; 11-20 Very large effect on the patient's life.
Time Frame: Days 3, 8, 15
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Clobex Lotion
Number analyzed (Participants) | 17 | 17
participants
  Day 3 Score 0 -1 No effect | 5 | 4
  Day 3 Score 2- 5 Small effect | 6 | 4
  Day 3 Score 6- 10 Moderate effect | 5 | 7
  Day 3 Score 11- 20 Very large effect | 0 | 2
  Day 8 Score 0 -1 No effect | 9 | 7
  Day 8 Score 2- 5 Small effect | 4 | 6
  Day 8 Score 6- 10 Moderate effect | 3 | 3
  Day 8 Score 11- 20 Very large effect | 1 | 1
  Day 15 Score 0 -1 No effect | 11 | 10
  Day 15 Score 2- 5 Small effect | 3 | 5
  Day 15 Score 6- 10 Moderate effect | 2 | 1
  Day 15 Score 11- 20 Very large effect | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline through Day 15.
Arm/Group | Olux-E Foam | Clobex Lotion
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 2/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olux-E Foam (N=17) | Clobex Lotion (N=17)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hpertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.